CLINICAL TRIAL: NCT03803826
Title: Use of Cardiac Strains for Optimization of Cardiac Resynchronization Therapy in Non-Responders
Brief Title: Cardiac Strains for Optimization of CRT in Non-Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-STRAINS
Record Dates: First submitted 2018-12-20; First posted 2019-01-15 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Heart Failure
Keywords: cardiac resynchronization therapy; non-responders

STUDY DESIGN:
Intervention Model Description: Patients not responding to Cardiac Resynchronization Therapy-Defibrillators (CRT-D) after 3 months from implementation are randomly divided into control and intervention groups. Atrioventricular interval is adjusted so that E and A waves do not overlap, the interventricular interval iss subsequently optimized to yield maximum improvement of the sum of longitudinal+radial+circumferential strains. The left ventricular ejection fraction (LVEF) and NYHA (New York Heart Association Classification improvement 3 months after optimization are evaluated and the use of other strain combinations assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT-D re-programming (Experimental): The ineffective previously implanted CRT-D is reprogrammed under supervision of transthoracic echocardiography to:
  1. adjust the atrioventricular interval so that E and A waves do not overlap
  2. the interventricular interval is subsequently optimized to yield maximum improvement of the sum of longitudinal+radial+circumferential strains.
  Transthoracic echocardiography is performed prior to optimization and 3 months after optimization (i.e., 3 and 6 months after the CRT implantation) and and New York Heart Association Classification (NYHA Classification; total score range 1-4) is being determined in accordance with the standard NYHA methods re-programming of the interventricular interval
  Interventions: Device: CRT-D re-programming; Diagnostic Test: Trans-Thoracic Echocardiography
- Control Group (No Intervention): Only trans-thoracic echocardiography is performed during follow-ups at 3 and 6 months from CRT implantations performed and New York Heart Association Classification (NYHA Classification; total score range 1-4) is being determined in accordance with the standard NYHA methods

INTERVENTIONS:
Device: CRT-D re-programming — The previously implanted, ineffective CRT-D is reprogrammed under supervision of Trans-Thoracic Echocardiography (TTE) to:
  1. adjust the atrioventricular interval so that E and A waves do not overlap
  2. the interventricular interval is subsequently optimized to yield maximum improvement of the sum of longitudinal+radial+circumferential strains.
  Arms: CRT-D re-programming
Diagnostic Test: Trans-Thoracic Echocardiography — This intervention relates to the determination of strains and atrioventricular interval and supplies data for reprogramming the ineffective CRT-D
  Transthoracic echocardiography performed to determine the left ventricular ejection fraction as an outcome measure is not considered intervention here (as it is also performed in the control group and that would cause an error cross-referencing.
  Arms: CRT-D re-programming

SUMMARY:
The aim of this study is to investigate the possibility of optimizing the performance of CRT-D in non-responding patients through utilization of cardiac strain speckle tracking

DETAILED DESCRIPTION:
In approximately 30% of patients, cardiac resynchronization therapy (CRT) fails to lead to any improvement of the patients' status.

In this study, an investigation of a possible method of optimization through speckle tracking of cardiac strains is attempted.

Patients not responding to Cardiac Resynchronization Therapy-Defibrillators (CRT-D) after 3 months are randomly divided into control and intervention groups. Atrioventricular interval is adjusted so that E and A waves do not overlap and the interventricular interval subsequently optimized to yield maximum improvement of the sum of longitudinal+radial+circumferential strains. The left ventricular ejection fraction (LVEF) and NYHA (New York Heart Association Classification improvement 3 months after optimization are evaluated and use of other strain combinations assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic heart failure with NYHA III/IV, pharmacological treatment options exhausted, LVEF below 30%, and QRS duration over 130ms who did not respond to the implantation of CRT-D

Exclusion Criteria:

* Age below 18
* response to the original CRT implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the left ventricular ejection fraction | 6 months from CRT-D implantation, 3 months from optimization
  Left ventricular ejection fraction measured by transthoracic echocardiography prior to optimizing and during a follow-up examination three month after optimizing

SECONDARY OUTCOMES:
Change in NYHA Classification | 6 months from CRT-D implantation, 3 months from optimization
  NYHA (New York Heart Association Classification measured using the standard NYHA range I to IV - I being the best result, IV the worst) was evaluated using a standard NYHA questionnaire before optimization and 3 months after optimization during a follow-up examination

CONTACTS AND LOCATIONS:
Overall Officials: David Sipula, MUDr., Principal Investigator — University Hospital Ostrava, Dpt of Cardiovascular Diseases
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia